CLINICAL TRIAL: NCT03310229
Title: Pulmonary Hypertension in Haemodialysis Patients :Frequency and Risk Factors
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AMHerez, principal investigator, Assiut University
Other Study IDs: AssiutUn
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Hypertension
Keywords: cardiovascular complications
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — X-Rays

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: plain chest x-ray — the participants will be subjected to plain chest x-ray with other tools to help diagnose pulmonary hypertension in haemodialysis patients

SUMMARY:
High mortality rates due to cardiovascular disease in end-stage renal disease patients been described by epidemiological and clinical studies. It accounts for approximately 50 percent of deaths in dialysis patients. Although controversial, this may be due to the presence of excess vascular calcification particularly in the form of extensive coronary artery calcification which can be observed even in very young dialysis patients. It was suggested that abnormalities of the right ventricular function in patients with end-stage renal disease were largely due to pulmonary hypertension which usually develops secondary to pulmonary artery calcifications.

DETAILED DESCRIPTION:
Primary whose mechanisms are incompletely known, is another vascular disease entity recently described in chronic kidney disease particularly in patients undergoing haemodialysis. It corresponds to 5th subtype of World Symposium on Pulmonary Hypertension classification established in 2008 in Dana Point and updated in 2013 in Nice. Pulmonary hypertension is defined by Pulmonary arterial pressure mean ≥25 mm Hg at rest measured by right heart catheterization. Its pathophysiological mechanism is controversy maybe explained by vascular calcification, blood flow in arteriovenous fistula and fluid overload. Primary pulmonary hypertension is a major problem of haemodialysis patients because of its high prevalence, sometimes reaching 68% and by its significant morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* 80 haemodialsis patients aged from 18 to 60 years old
* 80 haemodialysis patients are on regular haemodialysis for more than one year

Exclusion Criteria:

* All patients with a high probability of secondary pulmonary hypertension, those with the following history: chronic obstructive pulmonary disease, pulmonary embolism congenital heart disease, heart failure, Bilharziasis plus active HIV infection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 80 subjects undergoing haemodialysis for more than one year will be subjected to some diagnostic tools to detect and know the frequency of pulmonary hypertension(PH) among those patients.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Measurement of pulmonary arterial pressure | Pulmonary arterial pressure can be measured for a participant using echocardiography in less than one hour
  The participants will be subjected to a trans-thoracic echocardiography to measure pulmonary arterial pressure to detect and know the frequency of pulmonary hypertension in our haemodialysis patients for adequate care and early treatment and to study its possible risk factors to decrease morbidity and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed abbass, Principal Investigator — Assiut University
Locations (1):
- Assiut uni, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simonneau G, Gatzoulis MA, Adatia I, Celermajer D, Denton C, Ghofrani A, Gomez Sanchez MA, Krishna Kumar R, Landzberg M, Machado RF, Olschewski H, Robbins IM, Souza R. Updated clinical classification of pulmonary hypertension. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D34-41. doi: 10.1016/j.jacc.2013.10.029. PMID 24355639
- [Background] Nitta K, Ogawa T. Vascular calcification in end-stage renal disease patients. Contrib Nephrol. 2015;185:156-67. doi: 10.1159/000380980. Epub 2015 May 19. PMID 26023025
- [Result] Li Z, Liu S, Liang X, Wang W, Fei H, Hu P, Chen Y, Xu L, Li R, Shi W. Pulmonary hypertension as an independent predictor of cardiovascular mortality and events in hemodialysis patients. Int Urol Nephrol. 2014 Jan;46(1):141-9. doi: 10.1007/s11255-013-0486-z. Epub 2013 Jun 21. PMID 23793619
- [Result] Stompor T. An overview of the pathophysiology of vascular calcification in chronic kidney disease. Perit Dial Int. 2007 Jun;27 Suppl 2:S215-22. PMID 17556308